CLINICAL TRIAL: NCT00533546
Title: Activated Protein C in Acute Stroke Trial
Acronym: APCAST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Curtis Benesch, Associate Professor of Neurology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 537; 5R01HL080107 (NIH); 5R01HL080107-05 (NIH)
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Stroke
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Protein C; drotrecogin alfa activated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tier One (Experimental): Participants will receive APC by intravenous injection, receiving 50% of dose as a bolus and the remainder as an infusion over one ho.
  Interventions: Drug: Activated Protein C

INTERVENTIONS:
Drug: Activated Protein C — Intravenous APC (10, 15, 22, 33, 50, and 75 mcg/kg) administered to patients with acute ischemic stroke within 0 - 9 hours of symptom onset
  Other Names: Xigris

SUMMARY:
The purpose of this research study is to determine the safety and learn more about the dose of Activated Protein C (APC) in reducing the damage from stroke.

DETAILED DESCRIPTION:
An ischemic stroke occurs when there is damage to the brain caused by blockage in the blood vessels supplying the brain. Approximately 500,000 people in the United States experience this type of stroke each year. The only approved treatment for acute stroke is to attempt to dissolve the blood clot using t-PA (tissue plasminogen activator). This treatment must be given within 3 hours of symptom onset and is associated with a risk of brain hemorrhage (bleeding in the brain) of about 6% (6 in 100 patients).

Activated Protein C (APC) is a protein in the blood that is important in dissolving blood clots and reducing inflammation. Studies in animals suggest that APC may also protect brain cells from injury caused by a stroke. We are doing this study to determine if giving APC to individuals who have had a stroke will be safe and will reduce the damage to brain cells caused by the stroke. APC is currently approved by the Food and Drug Administration (FDA) for use in patients with severe, life-threatening infections.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of acute ischemic stroke; acute ischemic stroke is defined as the sudden onset of a measurable neurological deficit presumably attributable to focal cerebral ischemia, and otherwise not attributable to ICH or other disease process
* Symptom onset within 0-9 hours of administration of study medication Stroke onset is defined as the time of first symptoms or signs of neurologic deficit. If the onset of symptoms/signs is unwitnessed, time of onset is presumed to be the last time the patient was observed to be intact
* Neurologic deficit on examination with NIHSS of greater than 4 and less than 23
* In women of childbearing potential, a negative urine pregnancy test prior to enrollment (to be confirmed later by serum test)
* Signed informed consent by subject or authorized representative

Exclusion Criteria:

* Computed tomography scan of the brain with evidence of intracranial hemorrhage or any finding not consistent with acute ischemic stroke as cause of presenting symptoms
* CT imaging demonstrating hypodensity more than 1/3 of MCA territory or mass effect
* Neurological (other than presenting stroke) or psychiatric condition that may affect the patient's functional status or that may interfere with the patient's assessment
* Clinically relevant pre-existing neurological deficit (historical modified Rankin score greater than 2 regardless of cause)
* Treatment with tissue plasminogen activator or other thrombolytic agent within 3 months, including treatment with tissue plasminogen activator for current stroke
* Need for treatment with anti-platelet agent or anticoagulant within 36 hours
* Previous stroke or serious head trauma within 3 months
* Major surgery within previous 14 days
* History of intracranial hemorrhage
* Rapidly improving or minor symptoms
* Symptoms suggestive of subarachnoid hemorrhage
* Gastrointestinal hemorrhage or urinary tract hemorrhage within previous 21 days
* Arterial puncture at noncompressible site within the previous 7 days
* Seizure at onset of stroke
* Use of oral anticoagulant medications at time of symptom onset or treatment with subcutaneous or intravenous heparin within previous 48 hours with elevated partial thromboplastin time
* INR values greater than 1.5
* Platelet count less than 100,000/μL
* Glucose concentration less than 40 mg/dL or greater than 400mg/dL
* Participation in another clinical trial within the last 30 days, or planned participation in another clinical trial
* Women who are currently breast-feeding
* Known resistance to activated Protein C (Factor V Leiden mutation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Benesch, MD, MPH, Study Chair — University of Rochester
Locations (9):
- United States (9):
  - University of California Irvine Medical Center, Orange, California
  - Loyola University Medical Center, Maywood, Illinois
  - Washington University--Barnes-Jewish Hospital, St Louis, Missouri
  - SUNY Downstate, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Palmetto Health Richland, Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period spanned the following dates: October 2007 through July 2010. Location of recruitment and enrollment was in the emergency department of approved sites for patients presenting with acute ischemic stroke. Of the 9 participating sites, 3 actively enrolled.
Pre-assignment Details: No patients were excluded after enrollment.
Groups:
- Intravenous APC 10 Microgram/kg Dose: Participants will receive APC by intravenous injection, receiving 50% of dose as a bolus and the remainder as an infusion over one hour.
  Activated Protein C : Intravenous APC (10 mcg/kg) administered to patients with acute ischemic stroke within 0 - 9 hours of symptom onset
Period: Overall Study
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intravenous APC 10 Microgram/kg Dose: Participants will receive APC by intravenous injection, receiving 50% of dose as a bolus and the remainder as an infusion over one hour.
  Activated Protein C : Intravenous APC (10, 15, 22, 33, 50, and 75 mcg/kg) administered to patients with acute ischemic stroke within 0 - 9 hours of symptom onset
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intracranial Hemorrhage
Description: Intracranial Hemorrhage (ICH):
  Fatal ICH: Death ascribed to ICH confirmed by autopsy or CT imaging. Major non-fatal ICH: Hemorrhage within brain parenchyma associated with neurological deterioration or evidence of subdural, epidural or intraventricular hemorrhage on CT imaging, with or without symptoms.
  Symptomatic ICH: Hemorrhage within the territory of qualifying infarction with neurological deterioration as measured by > 2 point increase in the National Institutes of Health Stroke Scale (NIHSS) from previous examination; hemorrhage in different vascular territory associated with new neurologic deficit. All symptomatic ICH will be defined as a major ICH.
  Asymptomatic ICH: Presence of hemorrhage within the territory of qualifying infarction without neurological deterioration ascribed to the hemorrhage or presence of hemorrhage within brain parenchyma outside the territory of qualifying infarction without new neurologic deficit (would not be considered a major ICH)
Time Frame: Measured within 36-48 hours of treatment
Population: All participants enrolled were analyzed.
Measure: Number; unit: participants
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Number analyzed (Participants) | 12
participants | 0

2. Secondary Outcome: Mean Modified Rankin Scale Score
Description: Measure of disability as determined by categorical assignment on modified Rankin Scale.. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intravenous APC 10 Microgram/kg Dose: Participants will receive APC by intravenous injection, receiving 50% of dose as a bolus and the remainder as an infusion over one hour.
  Activated Protein C: Intravenous APC (10, 15, 22, 33, 50, and 75 mcg/kg) administered to patients with acute ischemic stroke within 0 - 9 hours of symptom onset
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Number analyzed (Participants) | 12
units on a scale | 2.91 (1.58)

3. Secondary Outcome: Mean Barthel Index Score
Description: Measure of functional recovery using Barthel Index (range 0-100). The Barthel scale or Barthel ADL index is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing ADL and mobility with 10 points given to each variable for a total of 100 points. A higher number is associated with a greater likelihood of being able to live at home with a degree of independence following discharge from hospital. The ten variables addressed in the Barthel scale are:
  presence or absence of fecal incontinence presence or absence of urinary incontinence help needed with grooming help needed with toilet use help needed with feeding help needed with transfers (e.g. from chair to bed) help needed with walking help needed with dressing help needed with climbing stairs and help needed with bathing
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Number analyzed (Participants) | 12
units on a scale | 67.7 (34.2)

4. Secondary Outcome: National Institutes of Health Stroke Scale (NIHSS)
Description: The NIHSS is a measure of neurologic deficit on a scale of 0-42, with 0 being normal. The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. The 11 items are:
  Level of Consciousness Horizontal Eye Movement Visual field test Facial Palsy Motor Arm Motor Leg Limb Ataxia Sensory Language Speech Extinction and Inattention
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Number analyzed (Participants) | 12
units on a scale | 5.0 (4.2)

ADVERSE EVENTS:
Time Frame: 90 days following enrollment
Description: Serious Adverse Events were collected without regard to the specific Adverse Event Term.
Arm/Group | Intravenous APC 10 Microgram/kg Dose
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous APC 10 Microgram/kg Dose (N=12)
worsening of neurological symptoms (Nervous system disorders) | 3 (5) — Three subjects experienced neurological worsening based on an increase in the NIHSS. None of these events were attributed to study medication.
Hospitalization > 24 hours (General disorders) | 3 (3) — Subjects hospitalized for > 24 hours after discharge following incident event
death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous APC 10 Microgram/kg Dose (N=12)
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 3
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Cardiomegaly (Cardiac disorders) | 1
Oedema peripheral (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Hypoglycaemia (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye discharge (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral candidiasis (Gastrointestinal disorders) | 1
Oral fungal infection (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Catheter site pain (General disorders) | 1
Discomfort (General disorders) | 1
Implant site pain (General disorders) | 1
Lethargy (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 6
Cellulitis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Renal injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Blood cholesterol increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Electrocardiogram change (Investigations) | 1
Neurological examination abnormal (Investigations) | 1
Vibration test abnormal (Investigations) | 1
White blood cell count increased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Ketoacidosis (Metabolism and nutrition disorders) | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Contusion (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Skin and subcutaneous tissue disorders) | 1
Brain oedema (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Insomnia (Nervous system disorders) | 3
Muscle spasticity (Nervous system disorders) | 3
Neurological symptom (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Small cell lung cancer stage unspecified (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Gastrointestinal tube insertion (Surgical and medical procedures) | 3
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Study was terminated after completion of Tier One dosing level (n=12 subjects) due to lack of recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No